CLINICAL TRIAL: NCT05038657
Title: Atezolizumab in Patients With Urinary Tract Squamous Cell Carcinoma: a Single Arm, Open Label, Multicentre, Phase II Clinical Trial
Brief Title: Atezolizumab Immunotherapy, in Immunotherapy Naive Patients With Urinary Tract Squamous Cell Carcinoma (UTSCC).
Acronym: AURORA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Cancer Research UK (Other); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RHM
Record Dates: First submitted 2021-09-07; First posted 2021-09-09 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2021-09

CONDITIONS: Squamous Cell Carcinoma; Urinary Tract Cancer
MeSH Terms: conditions — Carcinoma, Squamous Cell; Urologic Neoplasms | interventions — atezolizumab; Therapeutics

STUDY DESIGN:
Intervention Model Description: This study uses a Simon's 2-Stage optimal design with best ORR (% with a confirmed partial or complete response by RECIST v1.1) at a minimum of 12 weeks from commencing treatment as the primary endpoint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab (Experimental): Treatment will consist of atezolizumab, by IV infusion, at a fixed dose of 1680 mg, every 28 days (day 1 of each cycle, +/- 3 days), for up to one year. Each participant will receive up to 13 doses in total.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Treatment will consist of atezolizumab, by IV infusion, at a fixed dose of 1680 mg, every 28 days (day 1 of each cycle, +/- 3 days), for up to one year. Each participant will receive up to 13 doses in total.
  Other Names: Treatment

SUMMARY:
Atezolizumab in patients with urinary tract squamous cell carcinoma: a single-arm, open-label, multicentre, phase II clinical trial

DETAILED DESCRIPTION:
AURORA is a phase II open-label trial of Atezolizumab in patients with urinary tract squamous cell carcinoma (UTSCC). UTSCC is the most common of the rare urinary tract cancer histologies, comprising 2.1-6.7% of urinary tract cancers overall. There are few data available to guide treatment decisions for UTSCC. The AURORA trial will test the hypothesis that PD-L1 inhibition with atezolizumab immunotherapy is clinically effective, tolerable and safe, in patients with urinary tract squamous cell carcinoma (UTSCC). Translational endpoints will aim to determine characteristics for responsiveness to this treatment. AURORA was developed on behalf of the International Rare Cancers Initiative (IRCI) and the National Cancer Research Institute Bladder and Renal Group.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically confirmed cancer of the urinary tract with squamous cell carcinoma histology and without any TCC component. Mixed non-TCC histology is allowed if squamous cell carcinoma is the predominant histology 2. Newly diagnosed or progressive measurable disease as defined by RECIST version 1.1. To be considered measurable (and to be designated as a target lesion), a lesion must not have been treated with prior radiotherapy or focal ablation techniques 3. Suitable, in the judgment of the local investigator, for treatment with atezolizumab, with palliative intent 4. Adequate haematologic and end-organ function within 28 days prior to the first study treatment including:

  1. Absolute neutrophil count ≥ 1.5 x109/L
  2. Platelet count ≥ 100 x109/L
  3. Haemoglobin ≥ 90 g/L
  4. Aspartate transaminase (AST), alanine transaminase (ALT), and alkaline phosphatase ≤ 2.5 times the institutional upper limit of normal (ULN)
  5. Total bilirubin ≤ 1.5 times ULN (or ≤ 3 ULN in patients with Gilbert's syndrome)
  6. Calculated creatinine clearance ≥ 20 mL/min (Cockcroft-Gault formula) 5. Up to one prior line of systemic chemotherapy for UTSCC 6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 7. Life expectancy ≥ 12 weeks 8. Representative formalin-fixed paraffin-embedded (FFPE) tumour sample with an associated linked-anonymised pathology report that is available for central use in translational studies 9. Able to comply with all trial procedures and processes 10. Aged 18 years or over 11. Provision of written informed consent

Exclusion Criteria:

1. Any component of TCC histology
2. Planned for treatment with curative intent
3. Prior systemic immunotherapy (prior intra-vesical treatments are allowed)
4. Major surgery within 30 days prior to enrolment
5. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
6. Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
7. Use of oral or IV steroids for 14 days prior to enrolment. Use of inhaled corticosteroids, physiologic replacement doses of glucocorticoids (i.e., for adrenal insufficiency), and mineralocorticoids (e.g., fludrocortisone) is allowed
8. Administration of a live or attenuated vaccine within 4 weeks prior to enrolment (COVID-19 vaccination is allowed)
9. Treatment with any other investigational agent within 4 weeks prior to enrolment
10. Coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, unstable arrhythmias, unstable angina or congestive cardiac failure (New York Heart Association ≥ grade 2) within 6 months prior to enrolment
11. Patients with known HIV infection or with active tuberculosis
12. Patients with known active hepatitis B virus (HBV; chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test) or hepatitis C. Patients with past HBV infection or resolved HBV infection (defined as the presence of hepatitis B core antibody and the absence of HBsAg) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA
13. Autoimmune disease including myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone or with controlled Type I diabetes mellitus on a stable dose of an insulin regimen are eligible for this study
14. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan. A history of radiation pneumonitis in the radiation field (fibrosis) is permitted
15. Prior allogeneic stem cell or solid organ transplant
16. Patients who are pregnant or breastfeeding
17. Patients of child-bearing potential who are not able to use a highly effective method of contraception (as detailed in section 3.6)
18. A recent or current other cancer. Current non-melanoma skin cancer, cervical carcinoma in situ, or localized prostate cancer not requiring current treatment are permissible, as is a history of a separate other malignancy having completed all active treatment ≥2 years previously

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Response to | 36 months
  To determine the clinical activity of atezolizumab in patients with incurable histologically confirmed, immunotherapy naïve UTSCC
  To determine the clinical activity of atezolizumab in patients with incurable histologically confirmed, immunotherapy naïve UTSCC

SECONDARY OUTCOMES:
Progression free survival | 36 months
  3. To determine the progression-free survival (PFS) of patients treated with atezolizumab in this clinical setting

CONTACTS AND LOCATIONS:
Overall Officials: Simon Crabb, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crabb S, Wickens R, Jane-Bibby S, Dunkley D, Lawrence M, Knight A, Jones R, Birtle A, Huddart R, Linch M, Martin J, Coleman A, Boukas K, Markham H, Griffiths G. Evaluating atezolizumab in patients with urinary tract squamous cell carcinoma (AURORA): study protocol for a single arm, open-label, multicentre, phase II clinical trial. BMC Cancer. 2023 Sep 19;23(1):885. doi: 10.1186/s12885-023-11397-x. PMID 37726695